CLINICAL TRIAL: NCT05516043
Title: A Retrospective, Observational, Multicenter, Study to Collect Clinical Safety and Performance Data of POLYTHESE® Vascular Prostheses
Brief Title: Safety and Performance of POLYTHESE® Vascular Prosthesis
Status: Completed | Type: Observational
Sponsor: Perouse Medical (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-PT-01
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Aneurysm Arterial; Peripheral Arterial Disease; Marfan Syndrome; Arterial Dissections; Ehlers-Danlos Syndrome
MeSH Terms: conditions — Peripheral Arterial Disease; Marfan Syndrome; Dissection, Blood Vessel; Ehlers-Danlos Syndrome | interventions — Drug Implants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Implantation with POLYTHESE® — thoracic vascular surgery, abdominal vascular surgery and peripheral vascular surgery

SUMMARY:
POLYTHESE® study is a retrospective, observational, multicentre, case series which examine short and long-term outcomes of using POLYTHESE®. This study will be done on Real World Data to describe the safety and performance of the device.

PMCF Study.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following inclusion criteria in order to be eligible for inclusion in the study:

- Patient has a minimum of 1-year post-operative follow-up data available, or complete data to death

Exclusion Criteria:

- none

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: all potential subjects who are appropriate for study inclusion, i.e. subjects implanted with POLYTHESE® for at least one year, or with complete data to death. As the study explores real world data, there is no exclusion criteria for subjects and all subjects with POLYTHESE® implanted for at least one year and have not objected to the collect of their data will be included in the study.
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-11-26 (Actual)

PRIMARY OUTCOMES:
Performance: Primary patency rate | 1 year
  Patency rate
Safety : Mortality rate | 30 days

SECONDARY OUTCOMES:
Procedural success rate | 5 years
  Ability to use with no need for replacement by another device and, Effective vascular flow restoration after procedure and, In case of aneurysm, exclusion of aneurysmal portion after procedure.
Primary patency rate | 5 years
  rate patency of the bypass graft without procedure or intervention of the conduit itself (except for occlusion)
Primary assisted patency rate | 5 years
  defined as rate patency of the bypass graft with or without procedure or intervention of the conduit itself (except for occlusion) after device implantation
Secondary patency | 5 years
  defined as rate patency of the bypass graft with or without procedure or intervention of the conduit itself for occlusion after device implantation
Device Failure | 5 years
  * Uncontrolled blood leakage from device
  * Loss of structural integrity, e.g. rupture and/or exaggerated dilation (> 50 %)
  * Occlusion of the device
  * Total or partial replacement of the device required
Mortality rate | 5 years
  freedom % from death
Limb salvage rate | 5 years
  defined as freedom % from target limb amputation
Adverse events | 5 years
  any documented adverse events, including anticipated and non-anticipated adverse events

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU CAEN, Caen
  - CHU de NANTES, Nantes
  - CHU La Pitié Salpétrière, Paris

DOCUMENTS (1):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT05516043/Prot_000.pdf